CLINICAL TRIAL: NCT04789564
Title: Predictors of Cardiovascular Magnetic Resonancerelated Parameters: Intramyocardial Hemorrhage, Microvascular Obstruction , Area at Risk and Strain Related Parameters, and Their Effects on Adverse Ventricular Remodeling and MACEs in STEMI Patients After Primary PCI
Brief Title: Predictive Value of Cardiovascular Magnetic Resonance Related Parameters in STEMI Patients After Primary PCI for Adverse Left Ventricular Remodeling and Major Adverse Cardiovascular Events
Status: Completed | Type: Observational
Sponsor: Qian geng (Other)
Responsible Party: Sponsor-Investigator, Qian geng, Clinical Professor, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: qgeng-2021-2-16
Record Dates: First submitted 2021-03-05; First posted 2021-03-09 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2021-03

CONDITIONS: Cardiovascular Diseases
Keywords: Intramyocardial Hemorrhage(IMH); Microvascular Obstruction(MVO); Area at Risk(AAR); CMR Related Strain; ST-segment elevation myocardial
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: cardiovascular magnetic resonance (CMR) — Testing CMR on patients of 7 days and 6 months after myocardial infarction

SUMMARY:
This study aim to investigate the predictive value of CMR parameters: infarct size (IS), intramyocardial hemorrhage, microvascular obstruction, area at risk and CMR derived strain parameters with the Major Adverse Cardiovascular Events (MACEs) and myocardial remodeling afterinfarction.

DETAILED DESCRIPTION:
Investigators will enroll 500 patients with STEMI after PCI who were admitted to the Chinese PLA General Hospital and other eight hospitals across China: Wuhan Asia Heart Hospital; the First People's Hospital of Yunlin; Chaoyang Hospital, Capital Medical University; Hainan Hospital of PLA General Hospital; the Second Affiliated Hospital of Nanchang University; the Second Hospital of Hebei Medical University; Guizhou Provincial People's Hospital; Affiliated Hospital of Zunyi Medical College between January 2014 and December 2019. CMR was performed at 7 days and 6 months after primary PCI to assess the final infarction size(IS), microvascular obstruction (MVO), intramyocardial hemorrhage(IMH), area at risk (AAR) and related strain parameters. All patients will be followed up by 5 years after adimission. Cardiovascular events concluded stroke, repeat revascularization, rehospitalization for acute heart failure, nonfatal myocardial infarction, and all cause death. All adverse clinical events as well as study end points were monitored and adjudicated by the independent event committee.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years.
2. clinically diagnosed ST-segment elevation myocardial infarction.
3. Intended to undergo emergency PCI.
4. Voluntary enrollment and signed informed consent form.

Exclusion Criteria:

1. undergoing revascularization (PCI or coronary artery bypass grafting (CABG)) within 6 months;
2. Pregnant and breastfeeding women;
3. Contraindications of CMR: implanted cardiac defibrillator (ICD), claustrophobia, allergy to gadolinium
4. Liver or kidney failure;
5. Malignant tumor;
6. Unconscious at present;
7. systolic blood pressure (SBP) less than 80 mmHg;
8. Patients with bundle branch or fascicular block, insufficient ECG data.
9. Patients with other significant abnormal signs, laboratory tests and clinical disease are unsuitable for participation in the study accessed by clinicians.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators will enroll 500 patients with STEMI after PCI who were admitted to the Chinese PLA General Hospital and other eight hospitals across China between January 2016 and January 2019. CMR was performed at 7 days and 6 months after primary PCI to assess the final infarction size, microvascular obstruction (MVO), area at risk (AAR) and related strain parameters. All patients will be followed up by 5 years after addimission index.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
MACEs | follow up in five years
  MACEs concluding All-cause mortality, stroke, repeat revascularization, rehospitalization for acute heart failure, nonfatal myocardial infarction

SECONDARY OUTCOMES:
Left ventricular remodeling | 6 month after PCI
  Increase of LVEDV >20%
Contrast-induced acute kidney injury | 48 to 72 hours after PCI
  25% or 0.5 mg/dl increase in serum creatinine

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Korosoglou G, Giusca S, Montenbruck M, Patel AR, Lapinskas T, Gotze C, Zieschang V, Al-Tabatabaee S, Pieske B, Florian A, Erley J, Katus HA, Kelle S, Steen H. Fast Strain-Encoded Cardiac Magnetic Resonance for Diagnostic Classification and Risk Stratification of Heart Failure Patients. JACC Cardiovasc Imaging. 2021 Jun;14(6):1177-1188. doi: 10.1016/j.jcmg.2020.10.024. Epub 2021 Jan 13. PMID 33454266
- [Background] Amier RP, Tijssen RYG, Teunissen PFA, Fernandez-Jimenez R, Pizarro G, Garcia-Lunar I, Bastante T, van de Ven PM, Beek AM, Smulders MW, Bekkers SCAM, van Royen N, Ibanez B, Nijveldt R. Predictors of Intramyocardial Hemorrhage After Reperfused ST-Segment Elevation Myocardial Infarction. J Am Heart Assoc. 2017 Aug 15;6(8):e005651. doi: 10.1161/JAHA.117.005651. PMID 28862937
- [Background] Kidambi A, Mather AN, Motwani M, Swoboda P, Uddin A, Greenwood JP, Plein S. The effect of microvascular obstruction and intramyocardial hemorrhage on contractile recovery in reperfused myocardial infarction: insights from cardiovascular magnetic resonance. J Cardiovasc Magn Reson. 2013 Jun 27;15(1):58. doi: 10.1186/1532-429X-15-58. PMID 23806080
- [Background] Durante A, Laricchia A, Benedetti G, Esposito A, Margonato A, Rimoldi O, De Cobelli F, Colombo A, Camici PG. Identification of High-Risk Patients After ST-Segment-Elevation Myocardial Infarction: Comparison Between Angiographic and Magnetic Resonance Parameters. Circ Cardiovasc Imaging. 2017 Jun;10(6):e005841. doi: 10.1161/CIRCIMAGING.116.005841. PMID 28592591
- [Background] Liang K, Nakou E, Del Buono MG, Montone RA, D'Amario D, Bucciarelli-Ducci C. The Role of Cardiac Magnetic Resonance in Myocardial Infarction and Non-obstructive Coronary Arteries. Front Cardiovasc Med. 2022 Jan 17;8:821067. doi: 10.3389/fcvm.2021.821067. eCollection 2021. PMID 35111833
- [Background] Jensch PJ, Stiermaier T, Reinstadler SJ, Feistritzer HJ, Desch S, Fuernau G, de Waha-Thiele S, Thiele H, Eitel I. Prognostic relevance of peri-infarct zone measured by cardiovascular magnetic resonance in patients with ST-segment elevation myocardial infarction. Int J Cardiol. 2022 Jan 15;347:83-88. doi: 10.1016/j.ijcard.2021.11.017. Epub 2021 Nov 10. PMID 34767896
- [Background] Scarsini R, Shanmuganathan M, De Maria GL, Borlotti A, Kotronias RA, Burrage MK, Terentes-Printzios D, Langrish J, Lucking A, Fahrni G, Cuculi F, Ribichini F, Choudhury RP, Kharbanda R, Ferreira VM, Channon KM, Banning AP; OxAMI Study Investigators. Coronary Microvascular Dysfunction Assessed by Pressure Wire and CMR After STEMI Predicts Long-Term Outcomes. JACC Cardiovasc Imaging. 2021 Oct;14(10):1948-1959. doi: 10.1016/j.jcmg.2021.02.023. Epub 2021 Apr 14. PMID 33865789
- [Background] Hamirani YS, Wong A, Kramer CM, Salerno M. Effect of microvascular obstruction and intramyocardial hemorrhage by CMR on LV remodeling and outcomes after myocardial infarction: a systematic review and meta-analysis. JACC Cardiovasc Imaging. 2014 Sep;7(9):940-52. doi: 10.1016/j.jcmg.2014.06.012. PMID 25212800
- [Background] Ganame J, Messalli G, Dymarkowski S, Rademakers FE, Desmet W, Van de Werf F, Bogaert J. Impact of myocardial haemorrhage on left ventricular function and remodelling in patients with reperfused acute myocardial infarction. Eur Heart J. 2009 Jun;30(12):1440-9. doi: 10.1093/eurheartj/ehp093. Epub 2009 Apr 3. PMID 19346229